CLINICAL TRIAL: NCT05268757
Title: Effect of Probiotics on Oral Homeostasis During Oral Hygiene Discontinuation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Deerland Probiotics and Enzymes (Unknown)
Responsible Party: Principal Investigator, Daniel Belstrøm, DDS, PhD, DDS, PhD, Dr. odont, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UCPH_01_006
Record Dates: First submitted 2022-02-24; First posted 2022-03-07 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: Double blinded randomized clinical trial with a test and placebo group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Computerized randomization only known to the principal investigator, who are not directly involved in data collection or data analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): In this group participants will receive probiotic supplements twice a day (morning and evening) for at period of 28 days (14 days with oral hygiene discontinuation followed by 14 days with regular oral care).
  Interventions: Behavioral: Oral hygiene discontinuation
- Placebo (Placebo Comparator): In this group participants will receiveplacebo twice a day (morning and evening) for at period of 28 days (14 days with oral hygiene discontinuation followed by 14 days with regular oral care).
  Interventions: Behavioral: Oral hygiene discontinuation

INTERVENTIONS:
Behavioral: Oral hygiene discontinuation — Oral hygiene discontinuation for 14 days followed by 14 days of regular oral care

SUMMARY:
The present study is a double-blinded randomized clinical trial with a duration of 28 days.

DETAILED DESCRIPTION:
The present study is a double-blinded randomized clinical trial with a duration of 28 days.

80 orally and systemically healthy participant will be allocated in the test (probiotic) and the control (placebo) group at baseline.

The intervention is oral hygiene discontinuation, which will be applied at baseline and continue through day 14, followed by 14 days with regular oral care.

Clinical measurements and sampling will be performed at baseline, day 14 and day 28

Primary endpoint: Changes in microbial composition.

Secondary endpoints: Changes in clinical and immunological parameters

ELIGIBILITY:
Inclusion Criteria:

- age > 18 yrs.

Exclusion Criteria:

* Presence of oral diseases i.e. gingivitis, periodontitis and dental caries
* Current smokers
* Any systemic diseases and current use of any medication with known effect on oral health
* Use of systemic antibiotics within the latest three months
* Age < 18 yrs., and age > 30 yrs.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in microbial composition in dental | Baseline vs. Day 14 and Day 28
  Changes in alpha and beta diversity of microbial composition

SECONDARY OUTCOMES:
Changes in clinical parameters | Baseline vs. Day 14 and Day 28
  Changes in levels of dental plaque and gingival inflammation

OTHER OUTCOMES:
Changes in salivary levels of inflammatory cytokines | Baseline vs. Day 14 and Day 28
  Changes in mean salivary levels of selected inflammatory cytokines

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Department of Odontology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No